CLINICAL TRIAL: NCT05889091
Title: The Safety of a Buried, Free Fat Flap to Reduce Neck Morbidity Following Cancer Treatment: A Pilot Study
Brief Title: A Study of the Use of Fat Flap Reconstruction to Reduce Neck Injury After Cancer Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-102
Record Dates: First submitted 2023-05-17; First posted 2023-06-05 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Free fat flap; Reconstruction; Quality of life; 23-102
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: This is a descriptive, single-arm pilot study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quality of life questionnaires (Experimental): After the Fat Flap Reconstruction at 6 months post-operatively, all patients will be asked to complete the selected patient reported outcomes instruments and to complete clinical assessment with either the Head and Neck Surgery (HNS) or Plastic & Reconstructing Surgery (PLA) care team. Range of Motion (ROM) measurements using a goniometer will be completed by a member of the HNS clinical team. At 12 months post-operatively, all patients will be asked to complete the selected patient reported outcomes instruments and to complete clinical assessment. Patients will be asked to complete inter-incisor distance measurement and barium swallow assessment, done by a member of the SLP team. Range of Motion (ROM) measurements using a goniometer will be completed by a member of the HNS clinical team.
  Interventions: Other: HRQOL instruments; Other: LENT SOMA instrument

INTERVENTIONS:
Other: HRQOL instruments — These instruments include Face Q for Appearance, Eating & drinking, Swallowing, and Saliva (patient-reported); the Neck Dissection Impairment Index (patient-reported); the Long-term ENT-Subjective/Objective/Management/Analysis (LENT-SOMA) for skin-subcutaneous tissue, muscle-soft tissue, mucosa - oral and pharyngeal, salivary gland, and mandible (patient- and clinician-reported); modified barium swallow study (8-point penetration aspiration scale).
Other: LENT SOMA instrument — LENT SOMA instrument will also be provided to summarize objective quality-of-life-related measures recorded at 12 months postoperatively, including interincisor distance (mm); neck range of motion measured in degrees of flexion, extension, lateral flexion, and rotation to both sides; and shoulder range of motion, measured in degrees of abduction.

SUMMARY:
The purpose of this study is to find out whether the fat ALT flap procedure is a safe and practical option for reducing neck morbidity in HNSCC patients following cancer treatment of the neck. Neck morbidity after radiation therapy and surgery includes difficulty swallowing, neck or shoulder pain, stiffness, swelling, or changes to the appearance of the treated area. In addition, the researchers will find out whether the study procedure is effective at reducing neck morbidity and improving quality of life after cancer treatment. The researchers will measure quality of life by having participants answer questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Diagnosed with HNSCC (e.g., oropharyngeal, hypo/laryngeal SCC)
* Primary treatment is with radiotherapy with or without chemotherapy
* Salvage neck dissection is subsequently indicated for persistent or recurrent, nonmucosal disease in cervical lymph nodes
* At the time of salvage neck dissection additional flap coverage is indicated to improve carotid coverage or replace missing skin

Exclusion Criteria:

* Patients with primary site mucosal recurrence in addition to neck disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2026-05-16 (Estimated); Study Completion 2026-05-16 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that experience a complications | within 90 days post operatively
  Flap-related surgical complications - subjective and objective outcomes using validated instruments and CTCAE V5.0 i. Partial/total flap loss ii. Venous/arterial thrombosis iii. Infection iv. Hematoma v. Seroma Donor site i. Hematoma ii. Infection iii. Seroma iv. Dehiscence

SECONDARY OUTCOMES:
changes in HRQOL scores | 1 year
  Appearance scores in HNSCC patients is +/- 18.1 if a similar standard deviation is observed. For the Face-Q Eating & Drinking, the standard deviation is 22, corresponding to a half width of +/- 12.4. For the Face-Q Swallowing, the standard deviation is 26, corresponding to a half width of +/- 14.7. For the Face-Q Saliva, the standard deviation is 27, corresponding to a half width of +/- 15.3. Due to the small sample size of this study, examination of the HRQOL scores will be exploratory and hypothesis generating in nature.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Matros, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm